CLINICAL TRIAL: NCT06943326
Title: Effects of Enteral Nutrition Content on Disease Progression in Sepsis Patients
Status: Recruiting | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, HAKAN TOĞUÇ, Assistant professor, Inonu University
Other Study IDs: Inonu-NAD-HT-02
Record Dates: First submitted 2025-04-08; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Sepsis; Nutritional Deficiency
Keywords: sepsis; intensive care; nutrition
MeSH Terms: conditions — Sepsis; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: nutrition monitoring — There is no investigator intervention in the study. Patients' nutrition is recorded for one week from the beginning of the study.

SUMMARY:
The aim of this study was to investigate the effects of enteral nutrition content on disease progression in sepsis patients.

DETAILED DESCRIPTION:
Sepsis is a serious health problem with high mortality and morbidity rates worldwide. Over-activation of the inflammatory response and related organ dysfunctions are the main characteristics of sepsis. Rapid diagnosis and effective management are of vital importance in the treatment of sepsis. In this context, the role of enteral nutrition in the progression of the disease is increasingly being investigated.

Enteral nutrition is the practice of providing nutrients through the gastrointestinal tract and is a preferred method compared to parenteral nutrition in critical illnesses, especially in sepsis. The enteral route may reduce the risk of microbial translocation and modulate the immune system by maintaining intestinal integrity. Therefore, the content of enteral nutrition in sepsis patients may significantly affect the course of the disease.

Existing literature examines the effects of different enteral nutrient contents on patients with sepsis, with a particular focus on how macro- and micronutrient compositions can modulate inflammatory and immune responses. This study aims to examine the effects of enteral nutritional content on disease progression in patients with sepsis.

This prospective cross-sectional study will be conducted with patients diagnosed with sepsis being treated in the intensive care unit of Mehmet Akif Inan Training and Research Hospital. The study was planned to evaluate the effect of energy and nutrient intake on disease outcomes. Within the scope of the study, 60 patients diagnosed with sepsis will be followed up according to treatment in intensive care unit.

The inclusion criteria of the study include being diagnosed with sepsis and being 24 hours after the start of treatment in the intensive care unit and being able to receive enteral nutrition. Exclusion criteria included having chronic liver disease, chronic renal failure, active cancer disease and being on parenteral nutrition.

Data Collection General and health information of the participants will be obtained from the patient file. Nutritional information of the participants will be calculated by the researcher by noting the amount of food and formula taken with enteral nutrition for 7 days and 7-day food consumption will be calculated.

Biochemical and inflammatory data including glucose, albumin, CRP, haemoglobin, urea, creatinine, lymphocytes, leukocytes, monocytes, neutrophils, eosinophils, basophils will be obtained from the patient records at the beginning of the study and after 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with sepsis and being able to receive enteral nutrition 24 hours after starting treatment in the intensive care unit

Exclusion Criteria:

* chronic liver disease, chronic renal failure, active cancer or parenteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with sepsis who were older than 18 years and receiving enteral nutrition and receiving treatment in the Intensive Care Unit of Mehmet Akif Inan Training and Research Hospital were included.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Serum Glucose Level | Baseline and Day 7
  Change in fasting blood glucose level (mg/dL) from baseline to Day 7.
Change in Serum Albumin Level | Baseline and Day 7
  Change in serum albumin concentration (g/dL) from baseline to Day 7.
Change in Serum C-Reactive Protein (CRP) Level | Baseline and Day 7
  Change in serum CRP level (mg/L) from baseline to Day 7.
Change in Hemoglobin Level | Baseline and Day 7
  Change in hemoglobin concentration (g/dL) from baseline to Day 7.
Change in Serum Urea Level | Baseline and Day 7
  Change in serum urea concentration (g/dL) from baseline to Day 7.
Change in Serum Creatinine Level | Baseline and Day 7
  Change in serum creatinine concentration (g/dL) from baseline to Day 7.
Change in Absolute Lymphocyte Count | Baseline and Day 7
  Change in absolute lymphocyte count () from baseline to Day 7.
Change in Total Leukocyte Count | Baseline and Day 7
  Change in total leukocyte count (10^3/µL) from baseline to Day 7.
Change in Monocyte Count | Baseline and Day 7
  Change in absolute monocyte count (10^3/µL) from baseline to Day 7.
Change in Neutrophil Count | Baseline and Day 7
  Change in absolute neutrophil count (10^3/µL) from baseline to Day 7.
Change in Eosinophil Count | Baseline and Day 7
  Change in absolute eosinophil count (10^3/µL) from baseline to Day 7.
Change in Basophil Count | Baseline and Day 7
  Change in absolute basophil count (10^3/µL) from baseline to Day 7.

CONTACTS AND LOCATIONS:
Locations (1):
- Mehmet Akif Inan Training and Research Hospital, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data from participants were gathered solely for research objectives, adhering strictly to the ethical principles of confidentiality and protection. As such, it is not available for sharing.